CLINICAL TRIAL: NCT06688513
Title: Social Needs App for Oncology Patients Phase II
Acronym: SNAP-On II
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00422975; PD-S-0002-NIH-SBIR423 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2024-10-18; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Social Support (Formal and Informal); Mobile Application
Keywords: cancer; Social Support; Mobile Applications; Apps; Social Determinants of Health; SDH
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Let's Talk: Sharing information about Family Cancer Risk (Sham Comparator): Participants in the control group will complete questions about their SDH needs in the Carealth mobile app but will not have any helpful resources attached to it that meet these needs. Instead, as an attention control, control group participants will be sent to an interactive tool created and validated by the Centers for Disease Control called Let's Talk: Sharing Info About Your Family Cancer Risk. This is an interactive tool that patients can use to learn about how to talk with their family members about the family member's cancer risk.
  Interventions: Behavioral: Let's Talk: Sharing information about Family Cancer Risk
- Carealth App (Experimental): Participants in the treatment group will complete questions about their SDH needs in the Carealth app. Those with SDH needs will be referred to resources to meet those needs through Findhelp embedded into the app. Participants in the treatment group will complete this information pre-surgery, which will be considered a baseline measurement at the start of their participation in the trial. Participants in the treatment group will also receive reminders based on the post-surgery discharge instructions.
  Interventions: Device: Carealth Phone App

INTERVENTIONS:
Device: Carealth Phone App — The goal for this study is to assess Carealth app's ability to connect patients to resources to meet patient's identified SDH needs, with the end goal of assessing reduction in 30-day readmission and missed visits by connecting patients to resources to meet their social needs in a way that enables them to receive care earlier or avoid complications.
  Arms: Carealth App
Behavioral: Let's Talk: Sharing information about Family Cancer Risk — An interactive tool that patients can use to learn about how to talk with their family members about the family member's cancer risk
  Arms: Let's Talk: Sharing information about Family Cancer Risk

SUMMARY:
SNAP ON II is a two-arm, parallel-group, multi-center, randomized trial for patients diagnosed with cancer who are planning to undergo expected uncomplicated surgical intervention for their cancer. The study seeks to test whether a mobile app (developed by PistevoDecision) that identifies and connects patients to resources to meet their basic needs (e.g., housing, food, transportation, etc) ccan improve patient outcomes. Prior to their scheduled surgery, patients will download a mobile/web app that asks about their social needs. Then, the treatment group will be connected to community-based resources through FindHelp and the control group will receive access to the Centers for Disease Control tool called Lets Talk: Sharing Info About Your Family Cancer Risk.

DETAILED DESCRIPTION:
The goal for this study is to assess Carealth app's ability to connect patients to resources to meet patient's identified Social Determinant of Health (SDH) needs, with the end goal of assessing reduction in 30-day readmission and missed visits by connecting patients to resources to meet their social needs in a way that enables them to receive care earlier or avoid complications. Additionally, we will integrating the collection of SDH data with Electronic Health Record (EHR) data, per the initiatives from the Centers for Medicare and Medicaid Services (CMS), the US Office of the National Coordinator for Health Information Technology, and private EHR organizations.

The central hypothesis is that the access to resources in the Carealth app is associated with reduced 30-day readmission when compared to access to the sham app. To test this hypothesis, we will conduct a randomized clinical trial at multiple clinical sites. Our primary aim is to determine the proportion of 30-day readmission in the Carealth app group versus the sham app group. Further, we hypothesize that the time to SDH needs being met, time from oncologic consultation to surgery, and likelihood of missed/rescheduled appointments in the first 90-days post surgery will be reduced in the Carealth app group compared to the sham app. Thus, our secondary aim is to compare these outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* ECOG Performance Status11 score of 2 or less
* Diagnosed with cancer (e.g., head and neck; lung; breast; genitourinary; pancreatic; gastrointestinal; gynecological)
* Requires surgery, with an overnight stay in the hospital, as part of the treatment for their cancer.
* Surgery is considered low risk of major complication, as determined by the surgeon.
* Must be in one of the following categories: 1) have no evidence or suspicion of metastatic disease at time of consult, 2) metastatic in first-line treatment, or 3) metastatic with a 6-month or greater survival expectancy
* Not scheduled for surgery within 2 weeks
* Able to read and respond in English
* Have access to a smartphone, tablet, computer, or other device with an internet connection and web browser, ability and willingness to download the Carealth app
* Able to provide consent to the study

Exclusion Criteria:

* Diagnosis of cancers in the central nervous system, as these patients may experience cognitive function changes pre- or post-diagnosis that might influence their ability to use the app
* Diagnosis of cancers of the upper extremities, as they may experience limited physical function that may make it challenging to use a mobile app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
30-day Readmission post-surgery | 30 Days
Time to Social Determinants of Health Needs Addressed | 90 Days
  Time to event analysis of social determinants of health needs addressed from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Dean, ScD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Northwell Health Cancer Institute, Lake Success, New York
  - The University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
* Presentations at national scientific meetings: This will include scientific meetings where the content centers on SDHs. It will also include national meetings where content interest relates to cancer care and delivery care processes including the annual meetings of the American Society of Clinical Oncology.
  * Presentations at local conferences at Johns Hopkins University and other hospital partner sites: These will include departmental grand rounds and presentations at lecture series.
  * Presentations to local community groups focused on cancer patient needs, including patient advocacy groups associated with each partnering hospital.
  * We will also develop a tutorial session for presentation via webinars illustrating the technology and intended use, and final webinar presentations to the NCI Evaluation Panel.
Supporting Information: Study Protocol, SAP
Time Frame: Approximately 6 months after the end of the trial
Access Criteria: Undecided